CLINICAL TRIAL: NCT03123692
Title: A Randomised, Placebo-controlled, Blinded, Cross-over, Pilot Study to Explore Safety and Efficacy of NBMI Treatment of Patients With Mild, Moderate and Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: NBMI - Clinical Study on COPD
Acronym: Emera003COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EmeraMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Emera003
Record Dates: First submitted 2017-04-05; First posted 2017-04-21 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: COPD; COPD Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N,N'-Bis(2-mercaptoethyl)isophthalamide

STUDY DESIGN:
Intervention Model Description: A randomised, two arm, double-blind, placebo-controlled, cross-over, once daily for 14 days and 28 days follow up
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 14 days treatment with NBMI 300 mg/day
  Interventions: Drug: Emeramide
- Placebo (Placebo Comparator): 14 days treatment with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emeramide — Lipophilic, membrane passing Metal chelator and anti oxidant
  Other Names: NBMI; Irminix
  Arms: Treatment
Drug: Placebo — 14 days treatment with placebo
  Arms: Placebo

SUMMARY:
A pilot study to explore safety of the treatment with the antioxidant and metal chelator NBMI in COPD patients.

Investigational product: NBMI ((N1,N3-bis(2-mercaptoethyl) isophthalamide), INN: Emeramide

Indication: Mild, moderate and severe COPD with bronchitis

A randomised, two arm, double-blind, placebo-controlled, cross-over, once daily for 14 days pilot study in subjects with COPD with bronchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age between 45 and 75 years, including
2. Ex-smokers, who quit smoking > 6 months prior to screening visit, with a smoking history of at least 10 pack years
3. Diagnosis of COPD according to GOLD stages I-III, i.e. Post-beta-2-agonist FEV1/FVC < 0.70 and Post-beta-2-agonist FEV1 >30 % of predicted value
4. Active symptomatic COPD with a total COPD assessment test (CAT) score >10
5. Bronchitis with cough and sputum production during many days of the last month, and at least three months during the last year
6. Has signed informed consent for participation
7. Willingness and ability to comply with study procedures, visit schedules, and other instructions regarding the study.

Exclusion Criteria:

1. Patient with > 2 COPD exacerbation requiring treatment with systemic corticosteroids and/or antibiotics or hospitalization within the last year
2. Patient with COPD exacerbation requiring treatment with systemic corticosteroids and/or antibiotics or hospitalization within the last 4 weeks
3. New medication or change of dose for COPD treatment within 4 weeks prior to randomisation (chronic treatment with stable dose is allowed)
4. Ongoing treatment with systemic steroids, antibiotics, oxygen treatment, N-acetylcysteine (NAC) or roflumilast within 4 weeks of randomisation
5. Clinically significant heart failure, heart infarction, stroke or TIA within 12 months of study screening
6. Ongoing treatment with warfarin at screening visit
7. Ongoing treatment with medications that are metabolised or eliminated through the CYP P450 system, which could cause a drug interaction with the investigational product, as judged by the investigator, within 2 weeks of randomisation
8. Ongoing treatment with metal containing medications, such as iron supplement, lithium medications or antacids, within 2 weeks of randomisation
9. History of alcohol abuse or substance/drug abuse within 12 months prior to screening visit
10. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subjects at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
11. Any clinically significant abnormalities in clinical chemistry or haematology results at the time of screening, as judged by the investigator
12. Total alanine aminotransferase (ALT), aspartate aminotransferase (AST) or creatinine > upper limit of normal (ULN) at screening
13. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the investigator, including history of hypersensitivity to drugs with a similar chemical structure or class to NBMI
14. History of allergy/hypersensitivity to bisulphites (e.g. red/white wine)
15. Women of child bearing potential who do not consent to using acceptable methods of contraception (i.e. one of the following: combined hormonal contraception and progestogen-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability - Adverse events | 14 days
  To evaluate the safety and tolerability of NBMI daily oral administration for 14 days in patients with mild, moderate and severe COPD. Adverse events in terms of frequency and severity compared to placebo treatment.

SECONDARY OUTCOMES:
Cough - Changes from baseline in Leicester cough questionnaire compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on cough in patients with moderate and severe COPD. Changes from baseline in Leicester cough questionnaire compared to placebo treatment.
Individual symptoms CAT - Changes from baseline in COPD assessment (CAT) test compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on changes from baseline in COPD assessment (CAT) test compared to placebo treatment.
Individual symptoms mMRC - Changes from baseline in modified Medical Research Council (mMRC) dyspnoea scale compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on changes from baseline in in modified Medical Research Council (mMRC) dyspnoea scale compared to placebo treatment
Individual symptoms 6 min walking test - Changes from baseline in 6 Minute walk test measurements compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on changes from baseline in 6 Minute walk test measurements compared to placebo treatment
Individual symptoms MDP - Changes from baseline in Multidimensional Dyspnoea Profile (MDP) compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on changes from baseline in Multidimensional Dyspnoea Profile (MDP) compared to placebo treatment
Laboratory - Changes from baseline of standard haematology and clinical chemistry laboratory analyses (e.g. blood, kidney, liver, infections) compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on changes from baseline of standard haematology and clinical chemistry laboratory analyses (e.g. blood, kidney, liver, infections) compared to placebo treatment
Vital signs - Changes from baseline of vital signs (incl. oxygen saturation (spO2), blood pressure, pulse, body weight) compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on changes from baseline of vital signs (incl. oxygen saturation (spO2), blood pressure, pulse, body weight) compared to placebo treatment
Lung function FEV - Changes from baseline in pre-, post-bronchodilator and FVC compared to placebo treatment. | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on lung function in patients with mild, moderate and severe COPD on changes from baseline in pre-, post-bronchodilator and FVC compared to placebo treatment.
Lung function St George - Changes from baseline in St George´s respiratory questionnaire compared to placebo treatment | 14 days
  To investigate the efficacy of NBMI daily oral administration for 14 days on lung function in patients with mild, moderate and severe COPD on changes from baseline in St George´s respiratory questionnaire compared to placebo treatment